CLINICAL TRIAL: NCT00105027
Title: The Standard Care vs. COrticosteroid for REtinal Vein Occlusion (SCORE) Study: Two Randomized Trials to Compare the Efficacy and Safety of Intravitreal Injection(s) of Triamcinolone Acetonide With Standard Care to Treat Macular Edema
Brief Title: The Standard Care vs. COrticosteroid for REtinal Vein Occlusion (SCORE) Study
Acronym: SCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: National Eye Institute (NEI) (NIH); Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-99; 5U10EY014351-05 (NIH); 5U10EY014404 (NIH); 5U10EY014352 (NIH)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Macular Edema, Cystoid; Retinal Vein Occlusion
Keywords: macular edema; central retinal vein occlusion (CRVO); branch retinal vein occlusion (BRVO)
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- CRVO Observation (Active Comparator)
  Interventions: Other: Standard Care
- CRVO 1 mg dose triamcinolone acetonide (Active Comparator)
  Interventions: Drug: intravitreal triamcinolone injection
- CRVO 4 mg dose triamcinolone acetonide (Active Comparator)
  Interventions: Drug: intravitreal triamcinolone injection
- BRVO standard care (Active Comparator)
  Interventions: Other: Standard Care
- BRVO 1 mg dose triamcinolone acetonide (Active Comparator)
  Interventions: Drug: intravitreal triamcinolone injection
- BRVO 4 mg dose triamcinolone acetonide (Active Comparator)
  Interventions: Drug: intravitreal triamcinolone injection

INTERVENTIONS:
Other: Standard Care — CRVO: observation; BRVO: standard care
  Arms: BRVO standard care; CRVO Observation
Drug: intravitreal triamcinolone injection — 1 mg dose
  Arms: BRVO 1 mg dose triamcinolone acetonide; CRVO 1 mg dose triamcinolone acetonide
Drug: intravitreal triamcinolone injection — 4 mg
  Arms: BRVO 4 mg dose triamcinolone acetonide; CRVO 4 mg dose triamcinolone acetonide

SUMMARY:
The SCORE Study will compare the effectiveness and safety of standard care to intravitreal injection(s) of triamcinolone for treating macular edema (swelling of the central part of the retina) associated with central retinal vein occlusion (CRVO) and branch retinal vein occlusion (BRVO).

DETAILED DESCRIPTION:
Macular edema is a major cause of vision loss in patients with CRVO and BRVO. Both CRVO and BRVO are common retinal problems and are caused by a blockage in one of the large retinal veins (central retinal vein occlusion - CRVO) or smaller retinal veins (branch retinal vein occlusion - BRVO). Currently, there is no effective treatment for macular edema associated with CRVO and standard care treatment is observation. Grid laser photocoagulation may be effective for some patients for macular edema associated with BRVO, but many patients derive limited benefit from this treatment. Therefore, the development of new treatment modalities for macular edema caused by these two conditions is an important research goal.

Over the last several years, many patients with macular edema from CRVO and BRVO have been treated with an injection of a type of steroid called triamcinolone directly into the eye. This type of injection is called an intravitreal injection. The triamcinolone preparation commonly injected into the eye is Kenalog and is FDA-approved only for use in muscles and joints. The SCORE Study will use a formulation of triamcinolone made specifically for the eye.

The SCORE Study is a multicenter, randomized, Phase III trial to compare the effectiveness and safety of standard care versus triamcinolone injection(s) for the treatment of macular edema associated with CRVO and BRVO. In each of the two disease areas, 630 participants will be randomized (similar to a flip of a coin) in a 1:1:1 ratio to one of three groups: standard care, intravitreal triamcinolone 4 mg, or intravitreal triamcinolone 1 mg. After randomization, participants will be examined every 4 months through 3 years to collect ophthalmic information, including visual acuity, intraocular pressure, optical coherence tomography, and fundus photography . Fluorescein angiography will be performed at 4, 12 and 24 months. Repeat intravitreal injections of triamcinolone and repeat laser treatment will be provided as clinically indicated based on protocol-specific guidelines.

The primary outcome is improvement by 15 or more letters from baseline in best-corrected ETDRS visual acuity score at the 12-month visit. Secondary outcomes include changes from baseline in best-corrected ETDRS visual acuity score, changes in retinal thickness as assessed by stereoscopic color fundus photography and optical coherence tomography, and adverse ocular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with macular edema (swelling of the central part of the retina) associated with central retinal vein occlusion (CRVO) and branch retinal vein occlusion (BRVO).
* Individuals, 18 years of age or older, willing to provide consent may be eligible for the SCORE Study.

Exclusion Criteria: refer to SCORE Study website at https://web.emmes.com/study/score/ for listing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Ip, M.D., Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sets will be provided to qualified investigators under a Data Use Agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: to be set forth in data use agreement
Access Criteria: qualified investigators

REFERENCES:
- [Background] Bhavsar AR, Ip MS, Glassman AR; DRCRnet and the SCORE Study Groups. The risk of endophthalmitis following intravitreal triamcinolone injection in the DRCRnet and SCORE clinical trials. Am J Ophthalmol. 2007 Sep;144(3):454-6. doi: 10.1016/j.ajo.2007.04.011. PMID 17765429
- [Background] Scott IU, VanVeldhuisen PC, Oden NL, Ip MS, Blodi BA, Jumper JM, Figueroa M; SCORE Study Investigator Group. SCORE Study report 1: baseline associations between central retinal thickness and visual acuity in patients with retinal vein occlusion. Ophthalmology. 2009 Mar;116(3):504-12. doi: 10.1016/j.ophtha.2008.10.017. Epub 2009 Jan 22. PMID 19167078
- [Background] Scott IU, Blodi BA, Ip MS, Vanveldhuisen PC, Oden NL, Chan CK, Gonzalez V; SCORE Study Investigator Group. SCORE Study Report 2: Interobserver agreement between investigator and reading center classification of retinal vein occlusion type. Ophthalmology. 2009 Apr;116(4):756-61. doi: 10.1016/j.ophtha.2008.11.015. PMID 19344824
- [Background] Ip MS, Oden NL, Scott IU, VanVeldhuisen PC, Blodi BA, Figueroa M, Antoszyk A, Elman M; SCORE Study Investigator Group. SCORE Study report 3: study design and baseline characteristics. Ophthalmology. 2009 Sep;116(9):1770-1777.e1. doi: 10.1016/j.ophtha.2009.03.022. Epub 2009 Jul 19. PMID 19619896
- [Background] Domalpally A, Blodi BA, Scott IU, Ip MS, Oden NL, Lauer AK, VanVeldhuisen PC; SCORE Study Investigator Group. The Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) study system for evaluation of optical coherence tomograms: SCORE study report 4. Arch Ophthalmol. 2009 Nov;127(11):1461-7. doi: 10.1001/archophthalmol.2009.277. PMID 19901211
- [Background] Scott IU, Oden NL, VanVeldhuisen PC, Ip MS, Blodi BA, Antoszyk AN; SCORE Study Investigator Group. SCORE Study Report 7: incidence of intravitreal silicone oil droplets associated with staked-on vs luer cone syringe design. Am J Ophthalmol. 2009 Nov;148(5):725-732.e7. doi: 10.1016/j.ajo.2009.06.004. Epub 2009 Aug 11. PMID 19674727
- [Background] Oden N, Vanveldhuisen PC, Scott IU, Ip MS; the SCORE Study Investigator Group. SCORE Study Report 8: Closed Tests for All Pair-Wise Comparisons of Means. Drug Inf J. 2010 Jul 1;44(4):405-420. doi: 10.1177/009286151004400405. PMID 21660119
- [Background] Blodi BA, Domalpally A, Scott IU, Ip MS, Oden NL, Elledge J, Warren K, Altaweel MM, Kim JE, Van Veldhuisen PC; SCORE Study Research Group. Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) Study system for evaluation of stereoscopic color fundus photographs and fluorescein angiograms: SCORE Study Report 9. Arch Ophthalmol. 2010 Sep;128(9):1140-5. doi: 10.1001/archophthalmol.2010.193. PMID 20837797
- [Background] Scott IU, VanVeldhuisen PC, Oden NL, Ip MS, Blodi BA, Hartnett ME, Cohen G; Standard Care versus COrticosteroid for REtinal Vein Occlusion Study Investigator Group. Baseline predictors of visual acuity and retinal thickness outcomes in patients with retinal vein occlusion: Standard Care Versus COrticosteroid for REtinal Vein Occlusion Study report 10. Ophthalmology. 2011 Feb;118(2):345-52. doi: 10.1016/j.ophtha.2010.06.034. PMID 20926135
- [Background] Chan CK, Ip MS, Vanveldhuisen PC, Oden NL, Scott IU, Tolentino MJ, Blodi BA; SCORE Study Investigator Group. SCORE Study report #11: incidences of neovascular events in eyes with retinal vein occlusion. Ophthalmology. 2011 Jul;118(7):1364-72. doi: 10.1016/j.ophtha.2010.11.020. Epub 2011 Mar 26. PMID 21440942
- [Background] Domalpally A, Peng Q, Danis R, Blodi B, Scott IU, Ip M; SCORE Study Research Group. Association of outer retinal layer morphology with visual acuity in patients with retinal vein occlusion: SCORE Study Report 13. Eye (Lond). 2012 Jul;26(7):919-24. doi: 10.1038/eye.2012.59. Epub 2012 Apr 27. PMID 22538214
- [Result] Ip MS, Scott IU, VanVeldhuisen PC, Oden NL, Blodi BA, Fisher M, Singerman LJ, Tolentino M, Chan CK, Gonzalez VH; SCORE Study Research Group. A randomized trial comparing the efficacy and safety of intravitreal triamcinolone with observation to treat vision loss associated with macular edema secondary to central retinal vein occlusion: the Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) study report 5. Arch Ophthalmol. 2009 Sep;127(9):1101-14. doi: 10.1001/archophthalmol.2009.234. PMID 19752419
- [Result] Scott IU, Ip MS, VanVeldhuisen PC, Oden NL, Blodi BA, Fisher M, Chan CK, Gonzalez VH, Singerman LJ, Tolentino M; SCORE Study Research Group. A randomized trial comparing the efficacy and safety of intravitreal triamcinolone with standard care to treat vision loss associated with macular Edema secondary to branch retinal vein occlusion: the Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) study report 6. Arch Ophthalmol. 2009 Sep;127(9):1115-28. doi: 10.1001/archophthalmol.2009.233. PMID 19752420
- [Derived] Aref AA, Scott IU, Oden NL, Ip MS, Blodi BA, VanVeldhuisen PC; SCORE Study Investigator Group. Incidence, Risk Factors, and Timing of Elevated Intraocular Pressure After Intravitreal Triamcinolone Acetonide Injection for Macular Edema Secondary to Retinal Vein Occlusion: SCORE Study Report 15. JAMA Ophthalmol. 2015 Sep;133(9):1022-9. doi: 10.1001/jamaophthalmol.2015.1823. PMID 26086920
- [Derived] Scott IU, Vanveldhuisen PC, Oden NL, Ip MS, Domalpally A, Doft BH, Elman MJ, Blodi BA; SCORE Study Investigator Group. Baseline characteristics and response to treatment of participants with hemiretinal compared with branch retinal or central retinal vein occlusion in the standard care vs corticosteroid for retinal vein occlusion (SCORE) study: SCORE study report 14. Arch Ophthalmol. 2012 Dec;130(12):1517-24. doi: 10.1001/archophthalmol.2012.2728. PMID 23229691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 8, 2004, and February 29, 2008, 271 patients with central retinal vein occlusion (CRVO) were enrolled from 66 clinical sites and 411 patients with branch retinal vein occlusion (BRVO) were enrolled from 75 clinical sites across the United States.
  Participant flow data are reported for the primary outcome measure (12 months).
Groups:
- CRVO Observation: Standard care consists of observation of the macular edema.
- CRVO 1 mg Dose Triamcinolone Acetonide; BRVO 1 mg Dose Triamcinolone Acetonide: Treatment administered at baseline. At each 4-month visit during follow-up, the investigator assessed whether persistent or recurrent macular edema was present that warranted retreatment with the 1 mg dose. Patients and investigators were masked to the triamcinolone acetonide dose used (1 mg or 4 mg).
- CRVO 4 mg Dose Triamcinolone Acetonide; BRVO 4 mg Dose Triamcinolone Acetonide: Treatment administered at baseline. At each 4-month visit during follow-up, the investigator assessed whether persistent or recurrent macular edema was present that warranted retreatment with the 4 mg dose. Patients and investigators were masked to the triamcinolone acetonide dose used (1 mg or 4 mg).
- BRVO Standard Care: Standard care was observation followed by grid laser photocoagulation if and when clearing of the hemorrhage permits grid laser photocoagulation. For study eyes of BRVO participants without a dense macular hemorrhage at enrollment, standard care consisted of immediate grid laser photocoagulation. The determination of a dense hemorrhage in the center of the macula (and thus the timing of the grid laser photocoagulation) was left to the discretion of the investigator. At each 4-month visit during follow-up, the investigator assessed whether persistent or recurrent macular edema was present that warranted retreatment with the randomization assigned treatment. Only those eyes eligible for laser photocoagulation (i.e. eyes with BRVO and without a dense macular hemorrhage) were eligible for retreatment.
Period: Overall Study
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
Started | 88 | 92 | 91 | 137 | 136 | 138
Completed | 73 | 83 | 82 | 121 | 121 | 125
Not Completed | 15 | 9 | 9 | 16 | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide | Total
Number analyzed (Participants) | 88 | 92 | 91 | 137 | 136 | 138 | 682
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 35 | 34 | 62 | 54 | 55 | 265
  >=65 years | 63 | 57 | 57 | 75 | 82 | 83 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (12.8) | 67.4 (12.4) | 67.5 (12.0) | 66.9 (11.5) | 67.2 (11.5) | 68.1 (10.6) | 67.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 40 | 71 | 68 | 63 | 325
  Male | 48 | 49 | 51 | 66 | 68 | 75 | 357
Region of Enrollment [Number; unit: participants]
  United States | 88 | 92 | 91 | 137 | 136 | 138 | 682

OUTCOME MEASURES:

1. Primary Outcome: The Number of Study Participants Experiencing an Improvement by 15 or More Letters From Baseline in Best-corrected ETDRS Visual Acuity Score at the 12-month Visit
Description: Visual acuity testing was done using electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity testing at 3 meters using the Electronic Visual Acuity Tester by a SCORE certified technician. A masked visual acuity examiner with no knowledge of treatment assignments performed visual acuity testing at the 4-month, 12-month, 24-month and 36-month visits. An E-ETDRS visual acuity score of 85 is approximately 20/20, and a score of 20 letters is approximately 20/400. A visual acuity letter score change of 15 is about three lines on a vision chart.
Time Frame: Change from baseline to 12 months
Measure: Number; unit: Participants
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
Number analyzed (Participants) | 88 | 92 | 91 | 137 | 136 | 138
Participants | 5 | 22 [-6.4 to 4.1] | 21 [-6.3 to 4.0] | 35 [1.1 to 7.3] | 31 [2.8 to 8.6] | 34 [0.9 to 7.2]

2. Secondary Outcome: Changes From Baseline in Best-corrected ETDRS Visual Acuity Score
Time Frame: 12 months
Population: Participants who attended month 12 visit
Measure: Mean (95% Confidence Interval); unit: letters read
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
Number analyzed (Participants) | 73 | 83 | 82 | 121 | 121 | 125
letters read | -12.1 [-17.1 to -7.1] | -1.2 [-6.4 to 4.1] | -1.2 [-6.3 to 4.0] | 4.2 [1.1 to 7.3] | 5.7 [2.8 to 8.6] | 4.0 [0.9 to 7.2]

3. Secondary Outcome: Changes in Retinal Thickness as Assessed by Stereoscopic Color Fundus Photography and Optical Coherence Tomography
Time Frame: 12 months
Population: Participants who attended month 12 visit
Measure: Median (Inter-Quartile Range); unit: um
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
Number analyzed (Participants) | 68 | 72 | 78 | 120 | 113 | 112
um | -277 [-418 to -40] | -196 [-390 to -62] | -261 [-407 to -79] | -224 [-411 to -67] | -149 [-279 to -18] | -170 [-304 to -63]

4. Secondary Outcome: Adverse Ocular Outcomes
Time Frame: 12 months
Population: Participants experiencing an adverse event
Measure: Number; unit: events
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
Number analyzed (Participants) | 88 | 92 | 91 | 137 | 136 | 138
events
  Initiation of IOP-lowering medications | 7 | 18 | 32 | 3 | 11 | 57
  IOP > 35 mm HG | 1 | 5 | 8 | 1 | 2 | 14
  IOP > 10 mm HG above baseline | 2 | 15 | 24 | 1 | 12 | 50
  Laser peripheral iridotomy | 0 | 0 | 1 | 0 | 0 | 1
  Trabeculectomy | 0 | 0 | 0 | 0 | 0 | 0
  Tube shunt | 0 | 2 | 0 | 0 | 0 | 0
  Cataract: lens opacity onset or progression: number analyzed (Participants) | 66 | 77 | 76 | 115 | 110 | 110
  Cataract: lens opacity onset or progression | 12 | 20 | 25 | 15 | 27 | 38
  Cataract surgery | 0 | 0 | 4 | 3 | 0 | 4
  Infectious endophthalmitis | 0 | 0 | 0 | 0 | 0 | 1
  Noninfectious endophthalmitis | 0 | 0 | 0 | 0 | 0 | 0
  Retinal detachment | 0 | 0 | 0 | 1 | 1 | 0
  Iris neovascularization | 2 | 9 | 4 | 1 | 1 | 2
  Retinal neovascularization | 4 | 2 | 2 | 5 | 1 | 3
  Vitreous hemorrhage | 4 | 4 | 0 | 2 | 1 | 3
  YAG capsulotomy | 1 | 0 | 0 | 1 | 0 | 1
  Sector or panretinal photocagulation | 5 | 9 | 3 | 5 | 1 | 4
  Pars plana vitrectomy | 1 | 2 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Three years
Description: Clinical sites were required to report all adverse events via an electronic data capture system. Electronic forms designed to collect adverse event data were available for input at any time, including between scheduled visits.
Arm/Group | CRVO Observation | CRVO 1 mg Dose Triamcinolone Acetonide | CRVO 4 mg Dose Triamcinolone Acetonide | BRVO Standard Care | BRVO 1 mg Dose Triamcinolone Acetonide | BRVO 4 mg Dose Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/88 | 1/92 | 2/91 | 3/137 | 2/136 | 2/138
Serious Adverse Events (participants affected / at risk) | 32/88 | 37/92 | 53/91 | 47/137 | 49/136 | 79/138
Other Adverse Events (participants affected / at risk) | 76/88 | 87/92 | 89/91 | 118/137 | 132/136 | 133/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO Observation (N=88) | CRVO 1 mg Dose Triamcinolone Acetonide (N=92) | CRVO 4 mg Dose Triamcinolone Acetonide (N=91) | BRVO Standard Care (N=137) | BRVO 1 mg Dose Triamcinolone Acetonide (N=136) | BRVO 4 mg Dose Triamcinolone Acetonide (N=138)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anisometropia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anterior chamber disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Automatic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 5 (5) | 9 (10) | 28 (30) | 12 (16) | 16 (18) | 40 (46)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 12 (12)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 4 (5) | 3 (3) | 1 (1) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Choroidal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival filtering bleb leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticular hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Finger amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (4) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Iris neovascularisation (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic nerve cupping (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Polyp (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinopathy proliferative (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous prolapse (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO Observation (N=88) | CRVO 1 mg Dose Triamcinolone Acetonide (N=92) | CRVO 4 mg Dose Triamcinolone Acetonide (N=91) | BRVO Standard Care (N=137) | BRVO 1 mg Dose Triamcinolone Acetonide (N=136) | BRVO 4 mg Dose Triamcinolone Acetonide (N=138)
Blepharitis (Eye disorders) | 0 (0) | 3 (5) | 8 (19) | 4 (8) | 9 (16) | 6 (11)
Bronchitis (Infections and infestations) | 1 (1) | 3 (4) | 5 (6) | 5 (6) | 3 (3) | 4 (4)
Cataract (Eye disorders) | 10 (14) | 9 (12) | 14 (16) | 15 (27) | 19 (28) | 21 (25)
Cataract subcapsular (Eye disorders) | 3 (3) | 8 (8) | 12 (12) | 2 (3) | 13 (14) | 16 (18)
Conjunctival haemorrhage (Eye disorders) | 3 (7) | 34 (54) | 30 (57) | 9 (9) | 54 (88) | 54 (82)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 6 (6) | 4 (4)
Dry eye (Eye disorders) | 3 (6) | 3 (5) | 2 (3) | 5 (12) | 7 (13) | 6 (10)
Eye irritation (Eye disorders) | 2 (2) | 11 (12) | 9 (14) | 6 (8) | 17 (28) | 8 (9)
Eye pain (Eye disorders) | 6 (6) | 15 (25) | 18 (36) | 9 (13) | 23 (34) | 18 (26)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 6 (8) | 5 (7) | 0 (0) | 10 (11)
Foreign body in eye (Injury, poisoning and procedural complications) | 5 (5) | 31 (31) | 22 (22) | 4 (4) | 67 (67) | 31 (31)
Foreign body sensation in eyes (Eye disorders) | 4 (5) | 8 (8) | 3 (3) | 1 (1) | 13 (13) | 12 (14)
Glaucoma (Eye disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (3) | 1 (2) | 6 (7)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 7 (8) | 4 (4) | 4 (6) | 5 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 5 (5) | 4 (4) | 6 (6) | 6 (7)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 4 (4) | 6 (6) | 12 (12) | 12 (12)
Intraocular pressure increased (Investigations) | 8 (10) | 20 (24) | 42 (55) | 7 (9) | 19 (24) | 64 (88)
Iris neovascularisation (Eye disorders) | 2 (2) | 6 (7) | 3 (3) | 0 (0) | 2 (2) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 5 (6) | 4 (7) | 5 (8) | 5 (7) | 6 (7)
Macular oedema (Eye disorders) | 2 (2) | 6 (6) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Maculopathy (Eye disorders) | 5 (5) | 9 (10) | 10 (10) | 9 (10) | 12 (14) | 9 (10)
Myodesopsia (Eye disorders) | 8 (9) | 32 (44) | 34 (52) | 17 (23) | 59 (81) | 45 (64)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 6 (7) | 8 (8) | 5 (6) | 9 (10)
Photopsia (Eye disorders) | 3 (3) | 7 (8) | 4 (4) | 5 (6) | 10 (11) | 5 (6)
Retinal haemorrhage (Eye disorders) | 1 (1) | 6 (6) | 1 (2) | 4 (5) | 1 (1) | 2 (2)
Retinal neovascularisation (Eye disorders) | 6 (6) | 4 (4) | 6 (6) | 6 (8) | 1 (1) | 5 (5)
Retinal vascular disorder (Eye disorders) | 0 (0) | 6 (6) | 1 (2) | 2 (2) | 4 (4) | 3 (3)
Retinal vein occlusion (Eye disorders) | 4 (4) | 4 (4) | 3 (3) | 6 (6) | 3 (3) | 8 (10)
Vision blurred (Eye disorders) | 5 (6) | 6 (11) | 9 (13) | 14 (19) | 15 (19) | 17 (22)
Visual acuity reduced (Eye disorders) | 10 (10) | 12 (14) | 10 (15) | 6 (11) | 11 (12) | 13 (15)
Visual impairment (Eye disorders) | 5 (5) | 5 (5) | 3 (4) | 11 (14) | 9 (10) | 7 (10)
Vitreous detachment (Eye disorders) | 8 (9) | 16 (19) | 10 (12) | 15 (20) | 21 (25) | 12 (14)
Vitreous haemorrhage (Eye disorders) | 7 (7) | 8 (8) | 2 (2) | 2 (2) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2008-02-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT00105027/Prot_SAP_000.pdf
  • Informed Consent Form (2007-07-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT00105027/ICF_001.pdf